CLINICAL TRIAL: NCT01781741
Title: A Pilot Study of Stereotactic Body Radiation Therapy (SBRT) After TEMLA With or Without Minimally Invasive Surgery for Stage III and Stage IV (Oligometastatic) Non-small Cell Lung Cancer
Brief Title: Stereotactic Body Radiation Therapy After Surgery in Treating Patients With Stage III-IV Non-small Cell Lung Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 223812; NCI-2013-00055 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 223812 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (TEMLA and SBRT) (Experimental): Patients undergo TEMLA to remove the mediastinal lymph nodes followed by a single fraction of SBRT to the primary tumor (unless VATS procedure done) and mediastinal lymph node beds (if positive on TEMLA), with or without minimally invasive surgery.
  Interventions: Combination Product: therapeutic lymphadenectomy (TEMLA) and Stereotactic Body radiation therapy (SBRT); Other: quality-of-life assessment

INTERVENTIONS:
Combination Product: therapeutic lymphadenectomy (TEMLA) and Stereotactic Body radiation therapy (SBRT) — Undergo TEMLA and SBRT
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This pilot clinical trial studies stereotactic body radiation therapy after surgery in treating patients with stage III-IV non-small cell lung cancer. Stereotactic radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Lymphadenectomy may remove tumor cells that have spread to nearby lymph nodes in patients with non-small cell lung cancer. Giving stereotactic body radiation therapy after lymphadenectomy may kill any tumor cells that remain after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility/toxicity of combining transcervical extended mediastinal lymphadenectomy (TEMLA) with or without video-assisted thoracoscopic surgery (VATS) and stereotactic body radiation therapy (SBRT).

SECONDARY OBJECTIVES:

I. To assess time to initiation of chemotherapy following TEMLA with or without video-assisted thoracoscopic surgery (VATS)and SBRT.

II. To assess feasibility/toxicity of combining TEMLA with or without VATS and SBRT with various chemotherapy regimens (to be determined by medical oncologist based on patient and tumor characteristics).

III. To estimate survival following TEMLA with or without VATS and SBRT. IV. To define any differences in quality of life/toxicity following TEMLA with or without VATS and SBRT based on tumor location (peripheral/central).

V. To assess response for primary tumor control and overall survival in TEMLA only patients.

VI. To assess progression free survival for TEMLA with or without (VATS) patients.

OUTLINE:

Patients undergo TEMLA to remove the mediastinal lymph nodes followed by a single fraction of SBRT to the primary tumor (unless VATS procedure done) and mediastinal lymph node beds (if positive on TEMLA), with or without VATS.

After completion of study treatment, patients are followed up at 6,9, and 12 months, every 6 months for 2 years and annually for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Have histologically proven diagnosis of non-small cell lung cancer (NSCLC) (stage III and stage IV [to include limited volume metastases such as brain, bone, adrenal])
* Patients of child-bearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving and study related procedure
* Patients with chemotherapy prior to TEMLA are eligible

Exclusion Criteria:

* Contraindication to SBRT or TEMLA; this includes the inability to cooperate with any aspect of SBRT such as the inability to lie still and breathe reproducibly
* If patient has an open thoracotomy for lung cancer they will not be able to receive SBRT and will be replaced
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which the investigator's opinion deems the patient ineligible
* Received an investigational agent within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03-06 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Portion of patients with grade 3 or greater toxicity assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 4 | Up to 3 years
  Toxicity rates will be presented with Clopper-Pearson 90% confidence intervals.

SECONDARY OUTCOMES:
Time until chemotherapy | From the date of SBRT completion until the date of chemotherapy initiation, assessed up to 5 years
  A 90% confidence interval will be presented.
Incidence of toxicity associated with combining TEMLA with or without minimally invasive surgery stratified by chemotherapy regimens | Up to 5 years
  Exact 90% confidence intervals will be obtained for each unique chemotherapy regimen. Will be compared at each time-point between tumor locations using the Fisher's exact test.
Overall survival | From SBRT completion until death, assessed up to 5 years
  Will be described using standard Kaplan-Meier methodologies. The median survival time, 3-year survival rate, and 5-year survival rate and will be estimated and presented with 90% confidence intervals.
Quality of life (QoL) scores from European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 and EORTC QLQ Lung Cancer-Specific Module | Up to 5 years
  Will be compared with cumulative toxicity rates at each time-point between tumor locations using the Mann-Whitney U test. Comparisons of QoL scores between time-points will be made using the Wilcoxon signed rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

REFERENCES:
- [Derived] Singh AK, Hennon M, Ma SJ, Demmy TL, Picone A, Dexter EU, Nwogu C, Attwood K, Tan W, Hermann GM, Fung-Kee-Fung S, Malhotra HK, Yendamuri S, Gomez-Suescun JA. A pilot study of stereotactic body radiation therapy (SBRT) after surgery for stage III non-small cell lung cancer. BMC Cancer. 2018 Nov 29;18(1):1183. doi: 10.1186/s12885-018-5039-5. PMID 30497431